CLINICAL TRIAL: NCT05177003
Title: Study of the 12-month Efficacy of Stem Cell Injection in Crohn's Disease With Complex Ano-perineal Fistula
Acronym: ECESMAC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: ECESMAC
Record Dates: First submitted 2021-12-31; First posted 2022-01-04 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Crohn Disease; Ano Fistula
MeSH Terms: conditions — Crohn Disease; Rectal Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ano-perineal (or ano-rectal) fistulas are a frequent and major complication of Crohn's disease. Indeed, they indicate a greater severity of the disease. In addition, they have a major impact on the quality of life of patients. Finally, these fistulas are difficult to cure, especially when they are complex. Indeed, medical treatment with anti-TNF drugs can only cure them in one third of cases. Various obturation treatments have been proposed in addition to medical treatment such as advancement flap, injection of biological glue, placement of a plug, intersphincter ligation of the fistulous path or laser but with still insufficient healing rates.

The injection of mesenchymal stem cells of adipose origin was first proposed for this indication in 2003. Since then, numerous studies have been published on the subject. Most importantly, an international multicenter randomized double-blind phase 3 controlled trial demonstrated the superiority of allogeneic stem cells over placebo with a therapeutic effect maintained at one year follow-up. The trial involved selected patients with Crohn's disease and one or more complex ano-perineal fistulas refractory to conventional treatments. This treatment has a high cost and its practical modalities are constraining (manufacturing, delivery, constrained time between the factory and the injection). However, this study is the first to have demonstrated in such a rigorous way the effectiveness of a local treatment on complex ano-perineal fistulas of Crohn's disease. These allogeneic mesenchymal stem cells have therefore been granted marketing authorization in Europe and have been commercialized in several European countries including France during the summer of 2020 under the trade name ALOFISEL®. They are indicated for complex ano-perineal fistulas that have not responded to at least one conventional biological treatment, in the context of inactive or less active Crohn's disease.

The main objective of the study is to evaluate the rate of "deep" remission (i.e. clinical and radiological) at 12 months of follow-up in the first patients treated in France with ALOFISIEL® after its marketing. The evaluation is performed at 12 months because it seems that the result is consolidated after this period.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age ≥ 18 years
* Patient with inactive or minimally active Crohn's disease associated with one or more complex ano-perineal fistula(s) that has not responded to at least one conventional biologic therapy
* Patients managed for their fistula(s) by mesenchymal stem cell injection between July 1, 2020 and July 30, 2021 at one of the participating centers
* Patients who understand the French language

Exclusion Criteria:

* Patients under guardianship or curatorship
* Minor patients
* Pregnant women
* Patient deprived of liberty
* Patient under court protection
* Patients who object to the use of their data for this research
* Patients with a simple anal fistula
* Patients with anorecto-vaginal fistula
* Patients with anal canal stenosis that cannot be crossed by the index finger
* Patients who have not previously received medical treatment (biotherapy +/- immunosuppressant)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with inactive or minimally active Crohn's disease associated with one or more complex ano-perineal fistula(s) that has not responded to at least one conventional biologic therapy, managed for their fistula(s) by mesenchymal stem cell injection between July 1, 2020 and July 30, 2021 at one of the participating centers.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2021-07-02 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Deep remission rates | Month 12
  This outcome corresponds to the Rate of patients in deep remission at 12 months defined by the combination of:
  * absence of pain and oozing
  * closure of the secondary orifice(s) with the absence of discharge on digital pressure
  * absence of abscesses
  * absence of a collection of more than 20 mm on MRI.

SECONDARY OUTCOMES:
12-month clinical remission rate only | Month 12
  This outcome corresponds to the rate of patients in clinical remission alone at 12 months defined by the combination
  * an absence of pain and oozing
  * closure of the secondary orifice(s) with the absence of discharge on digital pressure
  * absence of abscesses
Primary clinical failure rate | Month 3
  This outcome corresponds to the rate of patients with primary treatment failure defined as non-closure of secondary orifice(s) with persistent flow on digital pressure at 3-month follow-up.
Evolution of the severity of the disease at 12 months | Month 12
  This outcome corresponds to the complication rates and types at 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia FATHALLAH, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (2):
- France (2):
  - Groupe Hospitalier Paris Saint-Joseph, Paris
  - CHU de Rennes, Rennes

REFERENCES:
- [Background] Alam A, Lin F, Fathallah N, Pommaret E, Aubert M, Lemarchand N, Abbes L, Spindler L, Portal A, de Parades V. FiLaC(R) and Crohn's disease perianal fistulas: a pilot study of 20 consecutive patients. Tech Coloproctol. 2020 Jan;24(1):75-78. doi: 10.1007/s10151-019-02134-3. Epub 2019 Dec 31. PMID 31893324
- [Background] Ciccocioppo R, Klersy C, Leffler DA, Rogers R, Bennett D, Corazza GR. Systematic review with meta-analysis: Safety and efficacy of local injections of mesenchymal stem cells in perianal fistulas. JGH Open. 2019 Feb 13;3(3):249-260. doi: 10.1002/jgh3.12141. eCollection 2019 Jun. PMID 31276044
- [Background] Garcia-Olmo D, Garcia-Arranz M, Garcia LG, Cuellar ES, Blanco IF, Prianes LA, Montes JA, Pinto FL, Marcos DH, Garcia-Sancho L. Autologous stem cell transplantation for treatment of rectovaginal fistula in perianal Crohn's disease: a new cell-based therapy. Int J Colorectal Dis. 2003 Sep;18(5):451-4. doi: 10.1007/s00384-003-0490-3. Epub 2003 May 20. PMID 12756590
- [Background] Mahadev S, Young JM, Selby W, Solomon MJ. Quality of life in perianal Crohn's disease: what do patients consider important? Dis Colon Rectum. 2011 May;54(5):579-85. doi: 10.1007/DCR.0b013e3182099d9e. PMID 21471759
- [Background] Panes J, Garcia-Olmo D, Van Assche G, Colombel JF, Reinisch W, Baumgart DC, Dignass A, Nachury M, Ferrante M, Kazemi-Shirazi L, Grimaud JC, de la Portilla F, Goldin E, Richard MP, Diez MC, Tagarro I, Leselbaum A, Danese S; ADMIRE CD Study Group Collaborators. Long-term Efficacy and Safety of Stem Cell Therapy (Cx601) for Complex Perianal Fistulas in Patients With Crohn's Disease. Gastroenterology. 2018 Apr;154(5):1334-1342.e4. doi: 10.1053/j.gastro.2017.12.020. Epub 2017 Dec 24. PMID 29277560
- [Background] Brochard C, Rabilloud ML, Hamonic S, Bajeux E, Pagenault M, Dabadie A, Gerfaud A, Viel JF, Tron I, Robaszkiewicz M, Bretagne JF, Siproudhis L, Bouguen G; Groupe ABERMAD. Natural History of Perianal Crohn's Disease: Long-term Follow-up of a Population-Based Cohort. Clin Gastroenterol Hepatol. 2022 Feb;20(2):e102-e110. doi: 10.1016/j.cgh.2020.12.024. Epub 2020 Dec 24. PMID 33359730
- [Background] Ford AC, Sandborn WJ, Khan KJ, Hanauer SB, Talley NJ, Moayyedi P. Efficacy of biological therapies in inflammatory bowel disease: systematic review and meta-analysis. Am J Gastroenterol. 2011 Apr;106(4):644-59, quiz 660. doi: 10.1038/ajg.2011.73. Epub 2011 Mar 15. PMID 21407183
- [Background] Stellingwerf ME, van Praag EM, Tozer PJ, Bemelman WA, Buskens CJ. Systematic review and meta-analysis of endorectal advancement flap and ligation of the intersphincteric fistula tract for cryptoglandular and Crohn's high perianal fistulas. BJS Open. 2019 Jan 21;3(3):231-241. doi: 10.1002/bjs5.50129. eCollection 2019 Jun. PMID 31183438
- [Background] Grimaud JC, Munoz-Bongrand N, Siproudhis L, Abramowitz L, Senejoux A, Vitton V, Gambiez L, Flourie B, Hebuterne X, Louis E, Coffin B, De Parades V, Savoye G, Soule JC, Bouhnik Y, Colombel JF, Contou JF, Francois Y, Mary JY, Lemann M; Groupe d'Etude Therapeutique des Affections Inflammatoires du Tube Digestif. Fibrin glue is effective healing perianal fistulas in patients with Crohn's disease. Gastroenterology. 2010 Jun;138(7):2275-81, 2281.e1. doi: 10.1053/j.gastro.2010.02.013. Epub 2010 Feb 20. PMID 20178792
- [Background] Senejoux A, Siproudhis L, Abramowitz L, Munoz-Bongrand N, Desseaux K, Bouguen G, Bourreille A, Dewit O, Stefanescu C, Vernier G, Louis E, Grimaud JC, Godart B, Savoye G, Hebuterne X, Bauer P, Nachury M, Laharie D, Chevret S, Bouhnik Y; Groupe d'Etude Therapeutique des Affections Inflammatoires du tube Digestif [GETAID]. Fistula Plug in Fistulising Ano-Perineal Crohn's Disease: a Randomised Controlled Trial. J Crohns Colitis. 2016 Feb;10(2):141-8. doi: 10.1093/ecco-jcc/jjv162. Epub 2015 Sep 8. PMID 26351393
- [Background] van Praag EM, Stellingwerf ME, van der Bilt JDW, Bemelman WA, Gecse KB, Buskens CJ. Ligation of the Intersphincteric Fistula Tract and Endorectal Advancement Flap for High Perianal Fistulas in Crohn's Disease: A Retrospective Cohort Study. J Crohns Colitis. 2020 Jul 9;14(6):757-763. doi: 10.1093/ecco-jcc/jjz181. PMID 31696918